CLINICAL TRIAL: NCT05073874
Title: Effects of Different Attentional Focus During Walking on Prefrontal Cortical Activation in Older Adults and Patients With Parkinson's Disease
Brief Title: Attentional Focus and Prefrontal Cortical Activation in Older Adults and Patients With Parkinson's Disease (PD)
Acronym: AttPark
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CHRO-2021-06
Record Dates: First submitted 2021-09-29; First posted 2021-10-12 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Parkinson Disease
Keywords: Attention; NIRS; Gait; Prefrontal cortex; Parkinson's disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Functional Near-Infrared Spectroscopy (fNIRS) (Other): Subjects will be guided to walk at a normal pace while maintaining the required attentional focus:
  1. no instructions about the attentional focus
  2. internal focus on their feet movements,
  3. external focus on two lines drawn on the floor,
  4. divided attention (walking while performing an arithmetic task).
  A fNIRS system will be used for the prefrontal cortex activation evaluation and connected soles for gait analyses.
  Interventions: Other: Functional Near-Infrared Spectroscopy (fNIRS)

INTERVENTIONS:
Other: Functional Near-Infrared Spectroscopy (fNIRS) — The hemodynamic response in prefrontal cortex will be measured using an Octomon+ system (Artinis). Eight emission and two detector probes will be arranged on the participant's forehead.

SUMMARY:
Attention may influence the motor performance and frontal activity. This study will examine the effect of different attentional focus: internal, external and divided attention (dual task) on prefrontal cortical activation (fNIRS) and on gait performance. Thirty older adults and thirty PD will participate in this study.

DETAILED DESCRIPTION:
The subjects will be guided to walk at a normal pace while maintaining the required attentional focus. Subjects will walk on 20 m four times in each of the four different focus conditions :

1. no instructions about the attentional focus
2. internal focus on their feet movements,
3. external focus on two lines drawn on the floor,
4. divided attention (walking while performing an arithmetic task).

A fNIRS system will be used for the prefrontal cortex activation evaluation and FeetMe soles for gait analyses.

ELIGIBILITY:
Inclusion Criteria:

* For 2 groups :

  * Man or woman 60-85 years old
  * Informed consent obtained
* Group Parkinson : clinical diagnosis of idiopathic Parkinson's Disease, according to the UK Brain Bank criteria.

Exclusion Criteria:

* For 2 groups :

  * Assisted walker
  * Neurological (other than those resulting from Parkinson's disease), cardiologic, rheumatologic disorders
  * Disorders affecting gait.
  * Montreal Cognitive Assessment (MOCA) < 24.
  * Concomitant medication likely to interfere with the results.
* Group Parkinson:

  * freezing
  * Hoehn et Yahr > III

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-12-08 (Actual); Primary Completion 2024-05-02 (Actual); Study Completion 2024-05-08 (Actual)

PRIMARY OUTCOMES:
Effects of oxyhemoglobin variations on hemodynamic response in prefrontal cortex | Baseline
  Oxyhemoglobin variations in prefrontal cortex will be measured with a fNIRS system, on a 20 meters distance.
Effects of deoxyhemoglobin variations on hemodynamic response in prefrontal cortex | Baseline
  Deoxyhemoglobin variations in prefrontal cortex will be measured with a fNIRS system

SECONDARY OUTCOMES:
Effects of speed on gait. | baseline
  Gait parameters will be measured with connected soles FeetMe ® : speed
Effects of cadence on gait. | baseline
  Gait parameters will be measured with connected soles FeetMe ® : cadence
Effects of stride length on gait. | baseline
  Gait parameters will be measured with connected soles FeetMe ® : stride length
Effects of double support time on gait. | baseline
  Gait parameters will be measured with connected soles FeetMe ® : double support time.

CONTACTS AND LOCATIONS:
Overall Officials: Canan OZSANCAK, Dr, Principal Investigator — CHR d'ORLEANS
Locations (1):
- CHR Orléans, Orléans, France

REFERENCES:
- [Background] Baltadjieva R, Giladi N, Gruendlinger L, Peretz C, Hausdorff JM. Marked alterations in the gait timing and rhythmicity of patients with de novo Parkinson's disease. Eur J Neurosci. 2006 Sep;24(6):1815-20. doi: 10.1111/j.1460-9568.2006.05033.x. PMID 17004944
- [Background] Hausdorff JM. Gait dynamics, fractals and falls: finding meaning in the stride-to-stride fluctuations of human walking. Hum Mov Sci. 2007 Aug;26(4):555-89. doi: 10.1016/j.humov.2007.05.003. Epub 2007 Jul 5. PMID 17618701
- [Background] Mahoney JR, Holtzer R, Izzetoglu M, Zemon V, Verghese J, Allali G. The role of prefrontal cortex during postural control in Parkinsonian syndromes a functional near-infrared spectroscopy study. Brain Res. 2016 Feb 15;1633:126-138. doi: 10.1016/j.brainres.2015.10.053. Epub 2015 Nov 6. PMID 26551767
- [Background] Plotnik M, Giladi N, Dagan Y, Hausdorff JM. Postural instability and fall risk in Parkinson's disease: impaired dual tasking, pacing, and bilateral coordination of gait during the "ON" medication state. Exp Brain Res. 2011 May;210(3-4):529-38. doi: 10.1007/s00221-011-2551-0. Epub 2011 Jan 30. PMID 21279632
- [Background] Yogev-Seligmann G, Rotem-Galili Y, Mirelman A, Dickstein R, Giladi N, Hausdorff JM. How does explicit prioritization alter walking during dual-task performance? Effects of age and sex on gait speed and variability. Phys Ther. 2010 Feb;90(2):177-86. doi: 10.2522/ptj.20090043. Epub 2009 Dec 18. PMID 20023000
- [Background] Pelicioni PHS, Tijsma M, Lord SR, Menant J. Prefrontal cortical activation measured by fNIRS during walking: effects of age, disease and secondary task. PeerJ. 2019 May 3;7:e6833. doi: 10.7717/peerj.6833. eCollection 2019. PMID 31110922
- [Background] Wulf G, Hoss M, Prinz W. Instructions for motor learning: differential effects of internal versus external focus of attention. J Mot Behav. 1998 Jun;30(2):169-79. doi: 10.1080/00222899809601334. PMID 20037032
- [Background] Holtzer R, Verghese J, Allali G, Izzetoglu M, Wang C, Mahoney JR. Neurological Gait Abnormalities Moderate the Functional Brain Signature of the Posture First Hypothesis. Brain Topogr. 2016 Mar;29(2):334-43. doi: 10.1007/s10548-015-0465-z. Epub 2015 Nov 27. PMID 26613725
- [Background] Maidan I, Bernad-Elazari H, Giladi N, Hausdorff JM, Mirelman A. When is Higher Level Cognitive Control Needed for Locomotor Tasks Among Patients with Parkinson's Disease? Brain Topogr. 2017 Jul;30(4):531-538. doi: 10.1007/s10548-017-0564-0. Epub 2017 Apr 24. PMID 28439757
- [Background] Yogev-Seligmann G, Hausdorff JM, Giladi N. The role of executive function and attention in gait. Mov Disord. 2008 Feb 15;23(3):329-42; quiz 472. doi: 10.1002/mds.21720. PMID 18058946
- [Background] Lu CF, Liu YC, Yang YR, Wu YT, Wang RY. Maintaining Gait Performance by Cortical Activation during Dual-Task Interference: A Functional Near-Infrared Spectroscopy Study. PLoS One. 2015 Jun 16;10(6):e0129390. doi: 10.1371/journal.pone.0129390. eCollection 2015. PMID 26079605
- [Background] Udina C, Avtzi S, Durduran T, Holtzer R, Rosso AL, Castellano-Tejedor C, Perez LM, Soto-Bagaria L, Inzitari M. Functional Near-Infrared Spectroscopy to Study Cerebral Hemodynamics in Older Adults During Cognitive and Motor Tasks: A Review. Front Aging Neurosci. 2020 Jan 21;11:367. doi: 10.3389/fnagi.2019.00367. eCollection 2019. PMID 32038224
- [Background] Kal EC, van der Kamp J, Houdijk H. External attentional focus enhances movement automatization: a comprehensive test of the constrained action hypothesis. Hum Mov Sci. 2013 Aug;32(4):527-39. doi: 10.1016/j.humov.2013.04.001. Epub 2013 Jun 30. PMID 24054892
- [Background] Nieuwhof F, Reelick MF, Maidan I, Mirelman A, Hausdorff JM, Olde Rikkert MG, Bloem BR, Muthalib M, Claassen JA. Measuring prefrontal cortical activity during dual task walking in patients with Parkinson's disease: feasibility of using a new portable fNIRS device. Pilot Feasibility Stud. 2016 Sep 23;2:59. doi: 10.1186/s40814-016-0099-2. eCollection 2016. PMID 27965875
- [Background] Yogev-Seligmann G, Sprecher E, Kodesh E. The Effect of External and Internal Focus of Attention on Gait Variability in Older Adults. J Mot Behav. 2017 Mar-Apr;49(2):179-184. doi: 10.1080/00222895.2016.1169983. Epub 2016 Aug 11. PMID 27715480
- [Background] Holtzer R, Mahoney JR, Izzetoglu M, Izzetoglu K, Onaral B, Verghese J. fNIRS study of walking and walking while talking in young and old individuals. J Gerontol A Biol Sci Med Sci. 2011 Aug;66(8):879-87. doi: 10.1093/gerona/glr068. Epub 2011 May 17. PMID 21593013
- [Background] Farid L, Jacobs D, Do Santos J, Simon O, Gracies JM, Hutin E. FeetMe(R) Monitor-connected insoles are a valid and reliable alternative for the evaluation of gait speed after stroke. Top Stroke Rehabil. 2021 Mar;28(2):127-134. doi: 10.1080/10749357.2020.1792717. Epub 2020 Jul 13. PMID 32654627